CLINICAL TRIAL: NCT02312427
Title: Investigation of the Impact of Dipeptidyl Peptidase-4 (DPP-4) Inhibition on Serum B-type Natriuretic Peptide (BNP) Level of Diabetic Patients With Congestive Heart Failure.
Brief Title: DPP-4 Inhibitor and Serum BNP Level of Diabetic Patients With Congestive Heart Failure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mitsui Memorial Hospital (Other)
Collaborators: Mitsukoshi Health and Welfare Foundation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MMHMEC2014-10
Record Dates: First submitted 2014-11-30; First posted 2014-12-09 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Heart Failure; Diabetes Mellitus
MeSH Terms: conditions — Heart Failure; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Outpatient arm (Experimental): After baseline data collection, DPP-4 inhibitor will be suspended for one month and serum BNP will be measured. The DPP-4 inhibitor will be resumed and after another month, serum BNP will be measured again.
  Interventions: Drug: Suspending DPP-4 inhibitor, in outpatient service
- Hospitalization arm 1 (Experimental): After hospitalization, medication for diabetes will be suspended. During the treatment for heart failure, drugs other than DPP-4 inhibitor will be resumed when required. After the stabilization of heart failure, DPP-4 inhibitor will be resumed (or administered if it was not prescribed before hospitalization) and serum BNP before and after the initiation of DPP-4 inhibitor will be measured.
  Interventions: Drug: Starting DPP-4 inhibitor after treatment of heart failure
- Hospitalization arm 2 (Experimental): After hospitalization, medication for diabetes may be suspended or continued. During the treatment for heart failure, drugs including DPP-4 inhibitor will be resumed when required. After the stabilization of heart failure, DPP-4 inhibitor will be suspended and serum BNP before and after the suspension of DPP-4 inhibitor will be measured.
  Interventions: Drug: Suspending DPP-4 inhibitor after treatment of heart failure

INTERVENTIONS:
Drug: Suspending DPP-4 inhibitor, in outpatient service — After baseline data collection, DPP-4 inhibitor (sitagliptin, vildagliptin, alogliptin, linagliptin, teneligliptin, anagliptin or saxagliptin) will be suspended for one month and serum BNP will be measured. The DPP-4 inhibitor will be resumed and after another month, serum BNP will be measured again.
  Arms: Outpatient arm
Drug: Starting DPP-4 inhibitor after treatment of heart failure — After hospitalization, medication for diabetes will be suspended. During the treatment for heart failure, drugs other than DPP-4 inhibitor will be resumed when required. After the stabilization of heart failure, DPP-4 inhibitor will be resumed (or administered if it was not prescribed before hospitalization) and serum BNP before and after the initiation of DPP-4 inhibitor will be measured.
  Arms: Hospitalization arm 1
Drug: Suspending DPP-4 inhibitor after treatment of heart failure — After hospitalization, medication for diabetes may be suspended or continued. During the treatment for heart failure, drugs including DPP-4 inhibitor will be resumed when required. After the stabilization of heart failure, DPP-4 inhibitor will be suspended and serum BNP before and after the suspension of DPP-4 inhibitor will be measured.
  Arms: Hospitalization arm 2

SUMMARY:
We thought to investigate the influence of DPP-4 inhibitor on the serum BNP level of diabetic patients with congestive heart failure. This study consists of two protocols. In the first protocol, diabetic patients with high level of serum BNP (100-2000 pg/ml) receiving outpatient treatment with any type of DPP-4 inhibitor at our institution will be enrolled. After baseline data collection, DPP-4 inhibitor will be suspended for one month and serum BNP will be measured. The DPP-4 inhibitor will be resumed and after another month, serum BNP will be measured again. In the other protocol, diabetic patients who were hospitalized due to heart failure were enrolled. DPP-4 inhibitor will be started (if the patient is not taking a DPP-4 inhibitor) or suspended (if the patient is taking a DPP-4 inhibitor) after stabilization of heart failure, and serum BNP will be measured before and after the drug administration or suspension.

ELIGIBILITY:
Outpatient arm

Inclusion Criteria:

* Type 2 diabetes patient with congestive heart failure under treatment with DPP-4 inhibitor (sitagliptin, vildagliptin, alogliptin, linagliptin, teneligliptin, anagliptin or saxagliptin) .
* High serum BNP (100-2000pg/ml).
* Patients who have given informed consent to participation in the study.

Exclusion Criteria:

* HbA1c over 9.0%.
* Patients who changed medication within 1 months before inclusion.
* Judged as ineligible by clinical investigators.

Hospitalization arm

Inclusion Criteria:

* Type 2 diabetes patient who were hospitalized for congestive heart failure.
* Patients who have given informed consent to participation in the study.

Exclusion Criteria:

* Patients on insulin therapy.
* Judged as ineligible by clinical investigators.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-01; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Serum BNP level with and without DPP-4 inhibitor use. | 3 days to 2 months
  In the outpatient arm, changes in serum BNP level measured 1 month after suspension of DPP-4 inhibitor, and 1month after resumption of the DPP-4 inhibitor will be analyzed. In the hospitalization arm, serum BNP before and 2-3 days after the initiation of DPP-4 inhibitor will be measured and compared.

SECONDARY OUTCOMES:
All cause mortality | 2 months
  Any deaths during the study period. (only for the outpatient arm)
Cardiovascular death | 2 months
  Any cardiovascular deaths during the study period. (only for the outpatient arm)
Heart failure hospitalization | 2 months
  Any hospitalization due to worsening of heart failure during suspension of or within 1month after resumption of taking a DPP-4 inhibitor. (only for the outpatient arm)
Worsening heart failure | 3 days
  Worsening of heart failure after the initiation of DPP-4 inhibitor. (only for the hospitalization arm)
Echocardiographic measures (Changes in echocardiographic measures during the study period.) | 3 days to 2 months
Other neurohormonal factors (Changes in plasma renin, aldosterone, serum stromal cell-derived factor 1 alpha, serum active glucagon-like peptide-1, serum active glucose-dependent insulinotropic polypeptid) | 3 days to 2 months
  Changes in plasma renin, aldosterone, serum stromal cell-derived factor 1 alpha, serum active glucagon-like peptide-1, serum active glucose-dependent insulinotropic polypeptide during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Akihiro Isogawa, M.D., Principal Investigator — Mitusui Memorial Hospital, Division of diabetes
Locations (1):
- Mitsui Memorial Hospital, Taito-ku, Tokyo, Japan